CLINICAL TRIAL: NCT01931215
Title: Transversus Abdominis Plane (TAP) Block Versus Intrathecal Morphine for Caesarean Section - Randomised Controlled Trial
Acronym: MOTAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benno Rehberg-Klug (Other)
Collaborators: Domitille Dereu (Unknown)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, Médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOTAP; CER 12-112 (Other: Comité d'éthique de la recherche des HUG)
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Ropivacaine; Clonidine

STUDY DESIGN:
Intervention Model Description: treatment versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: pharmacy providing identical sets of study drugs and placebo, computerized random sequence generation, sequence held by the pharmacy until study completion
Oversight: Data Monitoring Committee: No

ARMS (2):
- morphine group (Active Comparator): spinal anesthesia with intrathecal morphine
  Interventions: Other: spinal anesthesia with intrathecal morphine
- TAP group (Experimental): TAP-block with ropivacaine and clonidine
  Interventions: Other: TAP-block with ropivacaine and clonidine

INTERVENTIONS:
Other: spinal anesthesia with intrathecal morphine — in addition to the standard spinal anesthesia drugs (bupivacaine and fentanyl), morphine is added
  Arms: morphine group
Other: TAP-block with ropivacaine and clonidine
  Arms: TAP group

SUMMARY:
Analgesia after cesarean section is still not satisfactory for many women. Even if pain reduction is sufficient with the technique of intrathecal morphine injection, side effects such as nausea and pruritus are common.

Since several years, an alternative technique has been studied, the "transversus abdominis plane (TAP)"-block. Here a local anesthetic is injected in the abdominal wall muscles, and this has been shown to give a similar analgesic effect compared to intrathecal morphine, with potentially less side effects.

With this study, we want to evaluate if the TAP-block yields indeed less side effects when compared with intrathecal morphine.

The study will be a prospective study with the patients randomized to either a group with intrathecal morphine or a group with TAP-block.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be enrolled into the study:

* American Society of Anesthesiology (ASA) physical status less than 3 Able to read and understand the information sheet and to sign and date the consent form
* Scheduled for elective C-section planned with spinal anaesthesia
* Age>18

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

* Complicated pregnancy defined as having preeclampsia or placenta accreta, increta and percreta.
* Drug addiction.
* Contraindication to spinal anaesthesia (history of clotting disorders, septicemia, local infection at the injection site, spinal malformation, elevated intracranial pressure)
* Contraindication to TAP block (skin infection, abdominal wall muscle defect such as hernia and previous abdominal wall mesh).
* BMI>40 kg/m2
* Weight less than 50 kg the day of the C-section.
* Height less than 150 cm or more than 175 cm.
* Allergy/contraindication to any medication used in the study.
* Previous median abdominal incision. Necessity to perform the C-section urgently before the scheduled date (with less than 24h preparation time).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of nausea and/or vomiting at 24 hours | 24 hours
  Data for this endpoint will be gathered at 6h and 24h postoperatively from nurses' records in the recovery room (at 6h) and on the ward (at 24h), and counterchecked by asking the patient

SECONDARY OUTCOMES:
Cumulative incidence of pruritus at 24h | 24 h
  inquired directly from the patient at 6 and 24h
Cumulative incidence of treated nausea and vomiting at 24h | 24h
  (inquired directly from the patient at 6 and 24h).
Cumulative incidence of sedation at 6 and 24h. | 24h
  Sedation defined as an observer's assessment of alertness and sedation (OAAS) score lower than 4
Cumulative incidence of arterial hypotension | 24h
  defined as a systolic blood pressure of less than 100 mmHg for longer than 5 minutes (from nurse records at 6 and 24h)
Cumulative incidence of bradycardia | 24h
  defined as a heart rate of less than 50/min for longer than 5 minutes (from nurse records at 6 and 24h)
Cumulative incidence of respiratory depression | 24h
  defined as a respiratory frequency of less than 8/min for longer than 5 minutes (from nurse records at 6 and 24h
Cumulative morphine consumption at 24 hours | 24h
  (recorded in the memory of the patient controlled analgesia (PCA) pump).
Time until first PCA request | 24h
  (recorded in the memory of the PCA pump
Pain score at rest at 6, 24 and 48 hours postoperatively | 48h
  using the NRS scale (0-10)
Pain score on movement | 48h
  at 24 and 48 hours postoperatively (using the numerical rating scale (NRS 0-10)).
Maternal satisfaction at 24 and 48 hours postoperatively | 48h
  measured on a numeric rating scale (at 6h) and with the questionnaire "quality of recovery" (QoR40) at 24 and 48h
persistent pain at 3 and 6 months postoperatively | 6 months
  Pain at rest, 0-10 pain scale; Pain on movement, 0-10 pain scale; Yes/no for scar pain;Yes/no for analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Domitille Dereu, MD, Principal Investigator — HUG; Domitille Dereu, MD, Study Director — HUG
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Derived] Dereu D, Savoldelli GL, Mercier Y, Combescure C, Mathivon S, Rehberg B. The impact of a transversus abdominis plane block including clonidine vs. intrathecal morphine on nausea and vomiting after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2019 Aug;36(8):575-582. doi: 10.1097/EJA.0000000000001013. PMID 31274545